CLINICAL TRIAL: NCT06971718
Title: Drug Coated Balloons in Coronary Bifurcation Lesions. A Feasibility Study Looking at Computational Flow Dynamics, Ischaemic and Anatomical Changes to the Bifurcation
Brief Title: Coronary Bifurcations With Ischaemia and Flow Assessment
Status: Recruiting | Type: Observational
Sponsor: University of East Anglia (Other)
Collaborators: Norfolk and Norwich University Hospitals NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 325142
Record Dates: First submitted 2025-05-06; First posted 2025-05-14 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-04

CONDITIONS: Coronary Bifurcation Lesions
Keywords: Drug coated balloons; Coronary bifurcation lesions; Computational flow dynamics
MeSH Terms: interventions — Tomography, Optical Coherence

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Drug eluted stent
  Interventions: Diagnostic Test: Optical coherence tomography and pressure wire assessment of the vessel treated before and after treatment
- Drug coated balloon
  Interventions: Diagnostic Test: Optical coherence tomography and pressure wire assessment of the vessel treated before and after treatment

INTERVENTIONS:
Diagnostic Test: Optical coherence tomography and pressure wire assessment of the vessel treated before and after treatment — OCT and pressure wire of the main vessel and side branch of the bifurcation are undertaken prior to and after treating the lesion and at 3-9 month follow up.
  Other Names: Optical coherence tomography

SUMMARY:
The coronary arteries are blood vessels that provide oxygen rich blood to the muscle of the heart. If these vessels become narrowed or blocked, this can lead to chest pain (called angina) or heart attacks. Narrowings are usually treated using metal scaffolds called drug eluting stents. However, in one in five cases where the narrowing occurs at a branching point, treating it with stents is more challenging and can cause complications. A possible alternative treatment is using a special type of balloon called a drug-coated balloon. This balloon is inflated in the blood vessel and releases medicine to help widen the blood vessel and the procedure is completed without leaving any metallic scaffold behind.

This study aims to compare drug coated balloons with drug eluting stents to see which treatment works better for narrowing that occurs at branching points. We will used advanced imaging techniques to create computer models of blood flow in the vessels, and we will follow up with patients over tie to see how well the treatments work.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or over
* Any bifurcation lesion amenable to a provisional main vessel treatment strategy
* A main vessel diameter of 2.5mm or more and side branch diameter of >2mm
* Any patient with stable angina, silent ischaemia, unstable angina or NSTEMI
* Able to give informed consent

Exclusion Criteria:

* Cardiogenic shock
* LVEF <30%
* STEMI (as unable to give informed consent)
* eGFR <30
* Severe asthma contraindicating use of adenosine
* High degree AV block on 12 lead ECG precluding the use of adenosine
* Pregnancy
* Inability to consent
* Left main stem coronary bifurcation lesions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any patient with coronary bifurcation lesion who fulfills the inclusion criteria and is not precluded by the exclusion criteria is suitable for recruitment.
Sampling Method: Non-Probability Sample
Enrollment: 24 (Estimated)
Dates: Start 2023-10-10 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Physiological assessment | 3-9 months
  Physiological assessment measuring:
  * FFR (Main vessel and side branch)
  * Wall sheer stress
OCT derived anatomical measure | 3-9 months
  Mean lumen area main vessel and mean lumen area side branch

SECONDARY OUTCOMES:
Late lumen loss | 3-9 months
  Angiographic assessment of late lumen loss in main vessel and side branch
Device oriented clinical endpoints | 3-9 months
  Composite of:
  * Cardiovascular death
  * Device failure related MI
  * Device failure related ischaemia
  * Target bifurcation revascularisation
Patient focused endpoint: Angina | 12 months
  Seattle angina questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Vassilios S Vassiliou, Principal Investigator — Norwich Medical School; Simon C Eccleshall, Principal Investigator — Clinical Research and Trials Unit (Norfolk & Norwich University Hospital, UK)
Locations (1):
- Norwich Medical School, University of East Anglia, Norwich, Norfolk, United Kingdom

IPD SHARING:
Plan to Share IPD: No